CLINICAL TRIAL: NCT02620475
Title: A Randomized Split Scar Study of Suture Safe (South Medic) Treatment of Surgical Wounds to Minimize Scaring
Brief Title: A Randomized Split Scar Study of Suture Safe Treatment of Surgical Wounds to Minimize Scaring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: H15-02683
Record Dates: First submitted 2015-11-23; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Scars
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gold standard of care (Active Comparator): The usual gold standard of wound treatment to prevent scarring is to cover the incision with a self adhesive gauze type dressing (Mepore) covered by paper tape.
  Interventions: Device: SutureSafe
- SutureSafe dressings (Experimental): SutureSafe dressing are designed to apply a constant gentle inward pressure on the incision to reduce separating tension on newly formed incisions, stabilizing the healing environment.
  Interventions: Device: SutureSafe

INTERVENTIONS:
Device: SutureSafe — SutureSafe dressing are designed to apply a constant gentle inward pressure on the incision to reduce separating tension on newly formed incisions, stabilizing the healing environment.

SUMMARY:
The purpose of this study is to evaluate the effect SutureSafe dressings have on reducing scarring from an incision following an elective abdominoplasty (tummy tuck) procedure. The scar will be evaluated using subjective clinical assessment criteria. Each participant in the study will serve as a control and experiential study, since have of the incision will be treated with the gold standard of care and the other half with SutureSafe dressings.

DETAILED DESCRIPTION:
Patients of Dr. Nick Carr's who have elected to undergo an abdominoplasty (tummy tuck) procedure and have a fitzpatrick skin type of IV-VI will be offered participation in the study.

A full tummy tuck requires a horizontally-oriented incision in the area between the pubic hairline and belly button. The shape and length of the incision will be determined by the amount of excess skin. The excess skin is trimmed and the remaining skin is sutured together. A natural part of the healing process includes the body producing a fluid. The body is also able to reabsorb some fluid, but in the beginning there is more than the body can handle. Drains are inserted for one week post-operative to help remove that fluid. The usual standard of wound treatment to prevent scarring is to cover the incision with a self adhesive gauze type dressing (Mepore) covered by paper tape. The tape will be replaced at one-week post-operative and will be removed at two-weeks post-operative when the incision has fully healed. At this point the tape will then be replaced with a silicone strip for three additional months. In addition to the dressings the patient wearing a pressure garment for 1 month post-operative.

Patients who choose to be in the study, will have one half of the incision treated with the standard of care (explained in the previous paragraph) and the other side will be treated with SutureSafe dressings. Based on the Canadian medical device classification system, SutureSafe bandages are considered a class I device (which is the lowest risk category). The same process of wound care will be followed as outlined above, half of the incision will be treated with Mepore and paper tape, the other half of the incision will be treated with self-adhesive SutureSafe dressings. Both sides of the incisions will be replaced at one-week post-operative and will be removed at two-weeks post-operative when the incision has fully healed. At this point the tape will be replaced with a silicone strip and the SutureSafe bandages will be reapplied for three additional months.

The scar will be assessed at 3 months, 6 months and 1 year post-operative by observer Baillie Redfern. The clinical assessment of the scar will be performed using the Vancouver Scar Score criteria.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Have undergone an abdominoplasty procedure by Dr. Nick Carr
* Have fitzpatrick skin type IV-VI
* Be willing and able to return for all study follow-up procedures
* Have not participated in any other investigational or invasive clinical trial within the last 30 days, and will not participate in any other investigational or invasive clinical trial during this study; and
* Have been informed of the nature of the study, agreeing to its requirements, and have signed the informed consent approved by the Research Ethics Board.

Exclusion Criteria:

* Are unable to meet the treatment and follow up protocol requirements.
* Less than 18 years of ageCo-morbidity that reduces life expectancy to less than 12 months
* Cannot use any other methods (i.e. parmaceuditcal, natural, homeopathic) medications or devices for scar treatment.
* In the opinion of the Investigator, any medical condition that makes the subject unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change between usual standard of care and experimental dressings at 3 months, 6 months and 1 year, assessed using the Vancouver Scar Score | 3 months, 6 months and 1 year post operative

CONTACTS AND LOCATIONS:
Overall Officials: Nick Carr, B.Sc. MD, Principal Investigator — The University of British Columbia; Baillie L Redfern, B.Sc., M.Sc, Study Director — The University of British Columbia
Locations (1):
- Skin Works, Vancouver, British Columbia, Canada